CLINICAL TRIAL: NCT01120574
Title: Home Mechanical Ventilation in Patients With Chronic Obstructive Pulmonary Disease (COPD) Who Develop Nocturnal Hypercapnic Response Associated to Oxygen Therapy
Brief Title: Home Mechanical Ventilation in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Hypercapnic Response
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR05/05/2007
Record Dates: First submitted 2010-03-19; First posted 2010-05-11 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Nocturnal hypercapnic response to oxygen; Home mechanical ventilation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Oxygen therapy group.
- 2 (Active Comparator): Home mechanical ventilation plus oxygen therapy group.
  Interventions: Other: Home mechanical ventilation

INTERVENTIONS:
Other: Home mechanical ventilation — Home mechanical ventilation will be performed with a bilevel pressure ventilator.
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the clinical benefits of home mechanical ventilation associated to oxygen therapy in COPD patients with chronic respiratory failure (CRF) who develop hypercapnia and nocturnal respiratory acidosis secondary to oxygen administration.

We will include clinically stable COPD patients with hypercapnic CRF who develop a nocturnal hypercapnic response to oxygen (PaCO2 increase on awakening, at night with oxygen, >10 mmHg respect to PaCO2 breathing room air and awake). Obstructive sleep apnoea syndrome (OSAS) will previously have been excluded.

Patients will be admitted to the Pneumology ward where a nocturnal pulsioxymetry breathing oxygen therapy will be performed. Arterial blood gas samples will be taken at awakening (7AM).

Patients who develop a hypercapnic response to oxygen will be randomised into 2 treatment groups:

* Oxygen therapy group
* Home mechanical ventilation plus oxygen therapy group Home mechanical ventilation will be performed with a bilevel pressure ventilator. Functional respiratory variables as well as quality of life and sleep at onset and after 6 months treatment will be compared.

The principal outcome will be the evolution of arterial blood gases (PaCO2) between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients < 80 years old.
* COPD (ERS/ATS (FEV1 < 80%, FEV1/FVC < 70%, TLC > 80%)).
* Oxygen therapy indication (PaO2 < 55 mmHg or 55-59 associated to pulmonary arterial hypertension, chronic Cor Pulmonale, Chronic Heart failure, arrhythmias or polyglobulia).
* PaCO2 > 50 mm Hg.
* Clinically stable at least prior to one month.
* Hypercapnic response: increasing PaCO2 > 10 mmHg at 7 a.m after all night with oxygen compared with PaCO2 when awake and without oxygen therapy.

Exclusion Criteria:

* Active smoker.
* Bronchiectasis or tuberculous after-effects.
* Chronic respiratory failure secondary to thorax cage or neuromuscular diseases.
* BMI > 35 kg/m2
* OSAS.
* Locomotor system problems that disable 6 minutes walking test execution.
* Patients with tracheostomy.
* Other serious comorbidity (i.e chronic heart failure functional class > II NYHA, cancer or chronic renal failure that requires dialysis.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Arterial pressure of CO2. | Six months
  Follow up of its evolution comparing patients under O2 treatment and patients under O2 + non invasive ventilation treatment.

SECONDARY OUTCOMES:
Functional respiratory tests. | Six months
  Evolution during a follow up of 6 months between both groups (O2 vs O2+NIV).
Quality of life related to health | 6 months
  Evolution during a follow up of 6 months between both groups (O2 vs O2+NIV).
Nocturnal hypoventilation (nocturnal pulseoxymetry) | 6 months
  Evolution during a follow up of 6 months between both groups (O2 vs O2+NIV).

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Institu de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain